CLINICAL TRIAL: NCT05071521
Title: The Effectiveness of a Dissonance-based Eating Disorders Prevention Programme for Saudi Young Women
Brief Title: The Effectiveness of an Eating Disorders Prevention Program for Young Women in Saudi Arabia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PNU
Record Dates: First submitted 2021-09-17; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2020-10

CONDITIONS: Eating Disorder Symptom and Body Image Dissatisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eating disorders prevention (Active Comparator): The Body Project. The Body Project is a dissonance-based eating disorders prevention programme. It is a manualised evidence-based programme that targets eating pathology and body image dissatisfaction in young women. The objective of the programme is to create cognitive dissonance to encourage participants to decrease pursuing ideal-thinness. It includes group discussion, written and behavioural exercises and role-play to achieve cognitive dissonance (Stice, Rohde, & Shaw, 2013). It involves four group sessions for an hour each in consecutive weeks. At the beginning of each meeting, the facilitator reinforces voluntary commitment. Homework is explained and given at the end of each meeting and reviewed at the beginning of the following meeting.
  References:
  Stice, E., Rohde, P., Shaw, H. (2013). The body project a dissonance-based eating disorders prevention intervention (updated edition). New York: Oxford University Press.
  Interventions: Other: The Body Project: A Dissonance-Based Eating Disorder Prevention Intervention
- Healthy eating education (Sham Comparator): The control group were asked to read educational material in Arabic about healthy nutrition and active lifestyle from the Saudi branch of the World Obesity Federation (Kayl Association for Combatting Obesity, 2021). The material includes information about body mass index; easy ways to measure food units without a scale; benefits of working out; means to adopt healthier daily habits; and healthier food alternatives. The material was chosen because it was designed to be easy to understand by any individual.
  References:
  Kayl Association for Combatting Obesity. (2021). Kayl association for combatting obesity. Retrieved from https://www.kayl.org.sa
  Interventions: Other: The Body Project: A Dissonance-Based Eating Disorder Prevention Intervention

INTERVENTIONS:
Other: The Body Project: A Dissonance-Based Eating Disorder Prevention Intervention — The Body Project is a a selective dissonance-based prevention program that targets women with body image concerns. It has been developed with University and similar populations in mind, making it appropriate to the current research.The Body Project is based on a protocol, and aims to create cognitive dissonance that encourages participants to reduce pursuit of the thin-ideal. It involves the use of a scripted manual, covering four interactive weekly sessions. These involve role play, behavioural, verbal and written exercises.

SUMMARY:
The trial is a randomized control trial about the effective of an eating disorders prevention programmer for young Saudi women.

The prevention program is title The Body Project. Participants will be Saudi undergraduates from Princess Nourah Bint Abdulrahman University. Sample size is 64 participants. They will be divided randomly to two groups, each group has 32 participants. The first group is the intervention group where the prevention program will be provided. The second group will be the control group where healthy eating education material will be provided. The outcomes will be measured with adapted tools to local culture at three points (pre, post and 3 month follow-up).

ELIGIBILITY:
Inclusion Criteria:

undergraduate Saudi female

Exclusion Criteria:

undergraduate Saudi female with eating disorders

Ages: 16 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 92 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-07 (Actual); Study Completion 2021-03-07 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Examination-Questionnaire (EDE-Q, version 6.0). | 5 months
  The EDE-Q is a widely used self-report measure of eating disorder psychopathology (Fairburn & Beglin, 2008). It contains 28 items investigating eating disorder behaviours and attitudes during the past 28 days. It includes four subscales: dietary restraint; eating concerns; weight concerns; and shape concerns. The Global EDE-Q score (mean of the four attitudinal scores) and the scores of each subscales were used in this study. Higher scores indicate greater eating pathology. The scale was applied before and after the programme to assess outcomes.

SECONDARY OUTCOMES:
Body Shape Questionnaire (BSQ-8C). | 5 months
  Body image dissatisfactions was measured using the BSQ-8C, which is a short version of the full Body Shape Questionnaire (Evans & Dolan, 1993). A higher score indicates higher levels of body image dissatisfaction. The scale was applied before and after the programme to assess outcomes
Brief Version of the Fear of Negative Evaluation Scale (BFNE). | 5 months
  The BFNE (Leary, 1983) measures anxiety related to perceived negative evaluation. A high score shows higher levels of social anxiety. The scale was applied before and after the programme to assess outcomes.
Patient Health Questionnaire (PHQ-9). | 5 months
  Depression was assessed with the PHQ-9 (Löwe et al., 2004), which measures the severity of depression over the past two weeks. Higher scores indicate greater levels of depression. The scale was applied before and after the programme to assess outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Nourah Bint Abdulrahman University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided